CLINICAL TRIAL: NCT00299156
Title: Phase II Study of Oral Clofarabine in Myelodysplastic Syndrome (MDS)
Brief Title: Oral Clofarabine Study in Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0536
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-08

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic Syndrome; MDS; Chronic Myelomonocytic Leukemia; CMML; Clofarabine; Clofarex; Clolar; Chemotherapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Clofarabine (Experimental): 10 mg (Group 1) or 20 mg (Group 2) tablets once a day for 5 days in a row and repeated every 4-8 week cycle.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Starting dose 10 mg (Group 1) or 20 mg (Group 2) as tablets once a day for 5 days in a row and repeated every 4-8 weeks. Each 4-8 week period is a cycle.
  Other Names: Clolar®; Clorafex

SUMMARY:
The goal of this clinical research study is to learn if clofarabine given by mouth on a weekly schedule can help to control MDS. The safety of clofarabine given by mouth will also be studied.

DETAILED DESCRIPTION:
Clofarabine is a new chemotherapy drug that is designed to interfere with the growth and development of cancer cells.

If you are found to be eligible, you will be randomly assigned (as in the roll of dice) to one of 2 treatment groups. Participants in Group 1 will take a lower dose of clofarabine than Participants in Group 2. You have an equal chance of being assigned to either of the 2 treatment groups. Neither you nor your study doctor can choose your assignment. Later (after the first 40 patients), the assignment will favor the better treatment arm until one arm is selected as the significantly better one, or until 80 patients are treated in total. When you have been assigned to a treatment group, you will receive clofarabine as tablets once a day for 5 days in a row. This will be repeated every 4-8 weeks. Each 4-8 week period is considered 1 cycle of treatment.

Original patients who are still on study (original patients who received or are still receiving 30 mg/m2) have already been reduced to lower doses on subsequent courses or had treatment discontinued/completed. These patients will be asked to sign a new informed consent document to be made aware of the new developments in this study.

Each dose of clofarabine should be taken with 4 ounces of water in the morning, on an empty stomach. You must not eat or drink anything besides water from midnight the night before you take the study drug until 1 hour after taking the morning dose. You should take clofarabine every morning at about the same time. If vomiting occurs within 15 minutes of taking clofarabine, the dose may be repeated. If vomiting occurs more than 15 minutes after taking clofarabine, the dose cannot be replaced or made up.

Coffee and other caffeinated liquids cannot be taken before dosing and for 1 hour after dosing.

All clofarabine doses should be taken either in the outpatient or inpatient setting by qualified and trained site personnel or given with appropriate instructions to you and/or your care provider to take at home. At the start of each cycle, you will receive enough clofarabine for 1 cycle of therapy. You should store the clofarabine in its original container at room temperature. You should keep the container closed when not in use, and out of the reach of children.

After each cycle of therapy, you will not receive the next cycle of chemotherapy until your blood counts have recovered and any possible side effects have gone away (for around 4 to 8 weeks). You must stay in Houston for the first treatment cycle (about 4 to 8 weeks) and will be required to return to Houston before receiving each additional cycle of chemotherapy (up to 6 days each cycle).

Before every treatment cycle, your doctor will perform a physical exam, including measurement of your weight and vital signs (blood pressure, heart rate, temperature, and breathing rate). You will be asked about the level of your daily activities and how you are feeling. You will have blood samples (about 1-2 teaspoons) collected for routine lab tests 1-2 times a week for the first cycle, then every 2-4 weeks while on therapy. Repeat bone marrow samples will be collected every 1-3 cycles. However, if you complete the study before the third cycle, the bone marrow may be taken then. You may choose to have check-up visits and blood tests with your local doctor.

If you show a response and do not experience any severe side effects, you can receive up to a total of 12 cycles of therapy. During each cycle, clofarabine will be given the same way as during the first cycle. However, the dose of clofarabine may be lowered during later cycles to decrease the risk of side effects that may have occurred in previous cycles. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. Clofarabine given by vein is approved by the FDA for treatment of pediatric acute lymphoblastic leukemia. Its use in this study is experimental. Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS and >/= 5% blasts or IPSS risk intermediate or high; patients with Chronic myelomonocytic leukemia (CMML).
2. No prior intensive chemotherapy or high-dose ara-C (>/= 1g/m2).
3. Prior biologic therapies, targeted therapies, or single agent chemotherapy allowed.
4. Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease.
5. Hydroxyurea is permitted for control of counts prior to treatment.
6. Procrit, GCSF are allowed before therapy.
7. Performance 0-2 (ECOG). Adequate organ function including the following:Adequate liver function (bilirubin of < 2mg/dl), and renal function (creatinine < 2mg/dl), and SGPT (ALT) < 3 X ULN. Adequate cardiac functions (NYHA cardiac III-IV excluded).
8. Signed informed consent.

Exclusion Criteria:

1. Nursing and pregnant females. Patients of childbearing potential should practice effective methods of contraception. Child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Active and uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Prior clofarabine treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2006 to July 2012. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Sixty-five participants were registered, one participant did not receive study treatment. The study consisted of two parts, Phase 1 and a randomized Phase 2 portion.
Groups:
- Oral Clofarabine: Original dose of 40 mg oral reduced to 30mg and than lower dose of either 10 mg (Group 1) or 20 mg (Group 2) tablets once a day for 5 days in a row and repeated every 4-8 week cycle.
- Randomized, Oral Clofarabine 10mg: Arm A: 10 mg tablets once a day for 5 days in a row and repeated every 4-8 week cycle.
- Randomized, Oral Clofarabine 20mg: Arm B: 20 mg tablets once a day for 5 days in a row and repeated every 4-8 week cycle.
Period: Period 1 (Non-Randomized)
Arm/Group | Oral Clofarabine | Randomized, Oral Clofarabine 10mg | Randomized, Oral Clofarabine 20mg
Started | 32 | 0 | 0
Completed | 32 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2 (Randomized)
Arm/Group | Oral Clofarabine | Randomized, Oral Clofarabine 10mg | Randomized, Oral Clofarabine 20mg
Started | 0 | 17 | 16
Completed | 0 | 16 | 16
Not Completed | 0 | 1 | 0
Not completed — Screen Failure | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Clofarabine | Randomized, Oral Clofarabine 10mg | Randomized, Oral Clofarabine 20mg | Total
Number analyzed (Participants) | 32 | 17 | 16 | 65
Age, Continuous [Median (Full Range); unit: years] | 70.0 [53 to 86] | 67.5 [43 to 87] | 72.5 [54 to 84] | 70.0 [43 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 7 | 23
  Male | 23 | 10 | 9 | 42
Region of Enrollment [Number; unit: participants]
  United States | 32 | 17 | 16 | 65

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Complete Remission (CR)
Description: Complete Remission (CR): Normalization of the peripheral blood and bone marrow with <5% bone marrow blasts, a peripheral blood granulocyte count > (1.0 x 109/ L, and a platelet count > 100 x 109/L).
  Partial Remission: as above except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment.
  Hematologic Improvement: meets all criteria for CR except for platelet recovery to >100 x 109/L.
  Clinical Benefit: Platelets increase by 50% and to above 30 x 109/L untransfused (if lower than that pretherapy); or granulocytes increase by 100% and to above 109/L (if lower than that pretherapy); or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment > 5 x 109/L.
Time Frame: After 3 courses of treatment, up to 24 weeks.
Measure: Number; unit: Participants
Arm/Group | Oral Clofarabine | Randomized, Oral Clofarabine 10mg | Randomized, Oral Clofarabine 20mg
Number analyzed (Participants) | 32 | 16 | 16
Participants
  Complete Remission | 8 | 3 | 0
  Partial Remission | 0 | 0 | 0
  Hematologic Improvement | 3 | 1 | 3
  Clinical Benefit | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection with each 4-8 weeks course, up to a total of 12 courses of therapy. Overall study period, three years and four months.
Description: The first participant of the phase II portion of this study started treatment in August 2009.
Arm/Group | Oral Clofarabine | Randomized, Oral Clofarabine 10mg | Randomized, Oral Clofarabine 20mg
Serious Adverse Events (participants affected / at risk) | 16/32 | 8/16 | 12/16
Other Adverse Events (participants affected / at risk) | 32/32 | 16/16 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Clofarabine (N=32) | Randomized, Oral Clofarabine 10mg (N=16) | Randomized, Oral Clofarabine 20mg (N=16)
Death (General disorders) | 4 (4) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Death
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Tumor Lysis Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) — Death
Cerebrovascular Ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 7 (8) | 1 (1) | 3 (4)
Gastrointestinal Hemorrhage (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (1)
Vaginal Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 2 (2)
Fungal Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bone Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
E. Coli in Urine and Blood (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hemolytic Strep (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpetic Mouth Sores (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic Fever (Infections and infestations) | 0 (0) | 4 (6) | 7 (8)
Pseudomonas (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Clofarabine (N=32) | Randomized, Oral Clofarabine 10mg (N=16) | Randomized, Oral Clofarabine 20mg (N=16)
Fatigue (General disorders) | 15 (15) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (27) | 3 (3) | 6 (6)
Anorexia (Gastrointestinal disorders) | 7 (7) | 2 (2) | 1 (1)
Headache (General disorders) | 11 (11) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 0 (0) | 3 (3)
Abdominal Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated ALT (Metabolism and nutrition disorders) | 16 (16) | 1 (1) | 3 (3)
Elevated AST (Metabolism and nutrition disorders) | 22 (22) | 1 (1) | 1 (1)
Hyperbilirrubinemia (Metabolism and nutrition disorders) | 13 (13) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 8 (8) | 1 (1) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 5 (5) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1)
Musculoskeletal Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 18 (18) | 1 (1) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Alkaline Phosphatase (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 0 (0)
Palmoplantar Dysesthesia (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 0 (0)
Emesis (Gastrointestinal disorders) | 16 (16) | 0 (0) | 0 (0)
Gastrointestinal Hemorrhage (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Neutropenic Fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 16 (16) | 1 (1) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13) | 1 (1) | 1 (1)
Elevated Amylase (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes